CLINICAL TRIAL: NCT00615485
Title: Longitudinal Study of Bone Mineral Density in Survivors of Solid Pediatric Cancers
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Timothy Damron, M.D., Associate Professor, State University of New York - Upstate Medical University
Other Study IDs: Solid Pediatric Cancers; Joseph C. Georg Fund (Other: Sponsor name)
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Osteoporosis
Keywords: Examine the risk of osteoporosis in survivors of solid pediatric cancers
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — bone specific alkaline phosphatase n-telopeptide
Oversight: Data Monitoring Committee: No

SUMMARY:
Specific subgroups of children who survive treatment for childhood malignancies have been shown to develop relative osteopenia following chemotherapy and are felt to be at risk for developing osteoporosis later in life due to their inability to reach peak bone mass during childhood. Based upon an earlier study in our department, the investigators reported conclusive evidence that approximately half of survivors of pediatric solid malignancies are at risk for these problems. However, the proportion of patients in our population that showed osteopenia/osteoporosis was lower than that in other similar cross-sectional studies in solid tumors such as osteosarcoma. The main difference between our report and the osteosarcoma study was duration of follow-up, with ours being shorter. Longer follow-up may prove that a larger proportion of our patients are affected. The purpose is to perform a longitudinal follow-up study of bone mineral density using dual-energy X-ray absorptiometry (DXA) in adult survivors of solid pediatric tumors that were previously studied as subjects in our original cross-sectional study. The primary hypothesis is that the proportion of pediatric solid cancer survivors with significantly lower bone mineral density (BMD) compared to established age group controls will be increased with the additional time that has elapsed since the original study despite the fact that the patients are young and would not normally be expected to have osteopenia/osteoporosis at this age.

DETAILED DESCRIPTION:
AS ABOVE

ELIGIBILITY:
Inclusion criteria:

* The 38 patients from the SUNY Upstate Medical Center Pediatric Oncology Long-term Survivor Clinic who were subjects in the original Georg Fund supported study will comprise the patient population if they are locatable and willing to participate.
* Patients must be less than 40 years of age to participate.

Exclusion criteria:

* Patients who have received interval treatment for Acute Lymphocytic Leukemia (ALL) and those who have received subsequent cranial irradiation or total body irradiation (groups already known to be at high risk for osteoporosis) will be excluded. These would have had to have occurred in the interval since the original study, as these were also exclusion criteria for that study. In addition, any patient who received interval non-autologous bone marrow transplant will be excluded, as these patients may have graft versus host disease (also known to be associated with osteopenia).

Ages: 7 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The 38 patients from the SUNY Upstate Medical Center (Syracuse, NY) Pediatric Oncology Long-term Survivor Clinic who were subjects in the original Georg Fund supported study will comprise the patient population if they are locatable and willing to participate. Patients must be less than 40 years of age to participate.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2006-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Outcome Measure:pediatric solid tumor survivors are at an increased risk for developing generalized or regional osteoporosis as a result of chemotherapy for pediatric solid tumors. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A Damron, MD, Principal Investigator — SU
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States